CLINICAL TRIAL: NCT00547976
Title: PET Imaging of Peripheral Benzodiazepine Receptors in Patients With Carotid Atherosclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Robert B. Innis, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 080006; 08-M-0006
Record Dates: First submitted 2007-10-20; First posted 2007-10-23 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Atherosclerosis; Healthy
Keywords: Inflammation; Unstable Plaque; Macrophage; Thrombosis; Autoradiography; Atherosclerosis; Vasculitis
MeSH Terms: conditions — Atherosclerosis; Inflammation; Thrombosis; Vasculitis

INTERVENTIONS:
Drug: [C-11]PBR28

SUMMARY:
Inflammation in the vascular wall is important in atherosclerosis and the blockage of the artery. The peripheral benzodiazepine receptor is involved in inflammation and in this protocol we will attempt to take pictures, using PET camera, of inflammation in patients with atherosclerosis and compare those of healthy people.

DETAILED DESCRIPTION:
Objective

Inflammation in the vascular wall plays an important role in the pathophysiology of atherosclerosis, including development of plaque, plaque destabilization and rupture. Clinical and basic scientific data demonstrate the importance of peripheral white blood cells in this process. Therefore, a noninvasive method to detect inflammatory activity in atherosclerosis may be of great value to help determine prognosis, direct therapy and perhaps assess novel therapies for stabilization of atherosclerotic plaque.

The peripheral benzodiazepine receptor (PBR) is distinct from central benzodiazepine receptors associated with GABAA receptors and has been associated with immune function. PBR is expressed in macrophages, therefore, they may be a clinically useful marker to detect inflammation. Our preliminary autoradiographic data demonstrate specific PBR binding in carotid atherosclerosis samples. Though PBR has been imaged in vivo with positron emission tomography (PET) using [(11)C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195), we developed a new ligand, [(11)C]N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine (PBR28) that shows greater specific signal than [(11)C]PK11195 in non-human primates.

The objective of this protocol is to assess the utility of [(11)C]PBR28 PET to detect inflammation in unstable atherosclerosis plaques and large vessels with inflammation.

Study population

Twenty patients with carotid atherosclerosis, 20 patients with large vessel vasculitis including Takayasu's and Giant Cell arteritis, and 20 age-matched healthy subjects will have one PET scan.

Design

A [(11)C]PBR28 PET scan and a [18 F] fluorodeoxyglucose (FDG) PET scan will be performed in patients with carotid atherosclerosis. If the patient has endarterectomy after the PET scan, endarterectomy samples will be evaluated by in vitro autoradiography using [3H]PK 11195 and immunohistological staining with macrophage markers. Patients with large vessel vasculitis and healthy subjects will also have a [(11)C]PBR28 PET scan [18 F]FDG PET scan.

Outcome measures

Binding of [(11)C]PBR28 in atherosclerotic lesions, aortic arch and its branches will be compared with the binding in the contralateral carotid artery and those in healthy subjects. Binding of [(11)C]PBR28 will also be compared with accumulation of [18 F]FDG in each region. In addition, if the patients with atherosclerosis have endarterectomy, the binding in the atherosclerotic lesions will be compared with immunohistological staining of macrophage markers.

ELIGIBILITY:
* INCLUSION CRITERIA

Age 18 - 89

Ability to provide written informed consent

EXCLUSION CRITERIA

Severe systemic disease based on history, physical examination or laboratory tests that would prevent participation in the study

Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual guideline of RSC

Pregnancy and breast feeding

Claustrophobia

Inability to lie flat for a few hours for the PET scans

Medically unstable

The blood glucose level is greater than 150 mg/dL after fasting

Any other condition which in the opinion of the PI would prevent satisfactory participation in and completion of the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Binding of [11C]PBR28 at peripheral benzodiazepine receptor | 3 years

SECONDARY OUTCOMES:
PET [F-18]FDG uptake | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Anholt RR, Murphy KM, Mack GE, Snyder SH. Peripheral-type benzodiazepine receptors in the central nervous system: localization to olfactory nerves. J Neurosci. 1984 Feb;4(2):593-603. doi: 10.1523/JNEUROSCI.04-02-00593.1984. PMID 6321699
- [Background] Banati RB. Visualising microglial activation in vivo. Glia. 2002 Nov;40(2):206-217. doi: 10.1002/glia.10144. PMID 12379908
- [Derived] Schollhammer R, Lepreux S, Barthe N, Vimont D, Rullier A, Sibon I, Berard X, Zhang A, Kimura Y, Fujita M, Innis RB, Zanotti-Fregonara P, Morgat C. In vitro and pilot in vivo imaging of 18 kDa translocator protein (TSPO) in inflammatory vascular disease. EJNMMI Res. 2021 May 5;11(1):45. doi: 10.1186/s13550-021-00786-7. PMID 33950298